CLINICAL TRIAL: NCT01073241
Title: Transurethral Ventral Wall of Urethra-preserving Enucleation of Prostate
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Southwest Hospital, China (Other)
Responsible Party: JiHuixiang, Urology Department of Southwest Hospital, China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SouthwestH
Record Dates: First submitted 2010-02-22; First posted 2010-02-23 (Estimated); Last update posted 2010-03-15 (Estimated); Status verified 2010-02

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: benign prostatic hyperplasia; Transurethral Resection of Prostate; transurethral enucleation of prostate
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Transurethral Resection of Prostate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- transurethral prostatic resection (Active Comparator): The patients' prostate was resected with the conventional Nesbit TURP.
  Interventions: Procedure: transurethral prostatic resection
- ventral wall of urethra-preserving enucleation of prostate (Experimental): The patients' ventral wall of the prostate urethra was preserved and enucleation of prostate was performed for the left hyperplasia in the envelop.
  Interventions: Procedure: transurethral ventral wall of urethra-preserving enucleation of prostate

INTERVENTIONS:
Procedure: transurethral ventral wall of urethra-preserving enucleation of prostate — The patients' ventral wall of the prostate urethra was preserved and enucleation of prostate was performed for the left hyperplasia in the envelop.
  Other Names: TUEP
  Arms: ventral wall of urethra-preserving enucleation of prostate
Procedure: transurethral prostatic resection — The patients' prostate was resected with the conventional Nesbit TURP
  Other Names: TURP
  Arms: transurethral prostatic resection

SUMMARY:
In this study, the investigators designed a randomized and double-blind prospective trial to evaluate the efficiency and safety of the investigators new approach-transurethral ventral wall of urethra-preserving enucleation of prostate in comparison with TURP for the hyperplasia weighing more than 45 g.

DETAILED DESCRIPTION:
Although in recent dozen of years, laser operation and other safer minimally invasive surgeries have been well-developed, transurethral resection of the prostate (TURP) is still the gold standard for the surgical treatment of benign prostatic hyperplasia, despite of its various complications, and not suitable for the hyperplasia over 80 g which should be resected under open surgery. In this study, we design a randomized and double-blind prospective trial to evaluate the efficiency and safety of our new approach-transurethral ventral wall of urethra-preserving enucleation of prostate in comparison with TURP for the hyperplasia weighing more than 45 g.Urodynamic examination [maximum flow rate (QMax), detrusor pressure, and so on], transrectal color Doppler ultrasonography for the prostate, blood routine, blood electrolyte, prostate specific antigen (PSA), International Prostate Symptom Score (IPSS), the quality of life (Qol), blood loss during operation, and the weight of resected prostate were studied before and after the operation.

ELIGIBILITY:
Inclusion Criteria:

* BPH was diagnosed by DRE, Ultrasonography, CT or MR
* IPSS:>15
* Qmax:≤10ml/s and volume of bladder >200ml
* The weight of prostate >45g

Exclusion Criteria:

* Patient with other aggravating malignant tumor
* Total-PSA>20ng/ml, or 4<total-PSA<20ng/ml but the value of Free-PSA/total-PSA<0.16
* The maximum press of detrusor muscle <15cmH2O
* Patient with urethral stricture
* Patient with urinary infection
* Patient with Nervous System Disease
* Patient with surgical contraindication, such as severe cardiac or lung disease, diaphragmatic hernias, and so on

Ages: 45 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2010-03; Primary Completion 2012-02 (Estimated); Study Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
urodynamic study | before operation and the third month, 6th month after operation

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Jiahua, Study Director — Urology Institute of Southwest Hospital, Chongqin, China
Locations (1):
- Department of Urology, Southwest Hospital, Shapinba, Chongqin, China